CLINICAL TRIAL: NCT01903772
Title: Effects of Inspiratory Muscle Training in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: IMTCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Klaus Kenn, MD, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMTCO; Schön Klinik BGL (Other: Schön Klinik BGL)
Record Dates: First submitted 2013-07-12; First posted 2013-07-19 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: COPD; Inspiratory Muscle Weakness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory Muscle Training (Experimental): Procedure: Inspiratory Muscle Training Three times daily inspiratory muscle training (2x30 breaths) at an intensity of >50% Pi,max
  Interventions: Other: Inspiratory Muscle Training
- Sham Inspiratory Muscle Training (Sham Comparator): Twice daily inspiratory muscle training (3x30 breaths) at an intensity of 5 centimeters of water (H2O)
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training

SUMMARY:
The additional effect of inspiratory muscle training as an adjunct to a general exercise training program in patients with COPD with inspiratory muscle weakness will be studied. The main hypothesis is that inspiratory muscle training combined with an exercise training program improves functional exercise capacity more than an exercise training program without the addition of an inspiratory muscle training program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD
* Eligible to participate in an inpatient pulmonary rehabilitation program of 3 weeks
* Pi,max <60 centimeters of water or <50% of the predicted normal value

Exclusion Criteria:

* Major comorbidities preventing successful participation in an 8 week exercise training intervention
* use of non-invasive ventilation

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-04; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
6-Minute walking distance | change from the beginning at 3 weeks of a inpatient pulmonary rehabilitation program

SECONDARY OUTCOMES:
exercise capacity (constant work rate test) | change from the beginning at 3 weeks of a inpatient pulmonary rehabilitation program
maximal inspiratory pressure (PImax) | change from the beginning at 3 weeks of a inpatient pulmonary rehabilitation program
inspiratory muscle endurance capacity | change from the beginning at 3 weeks of a inpatient pulmonary rehabilitation program
dyspnea | change from the beginning at 3 weeks of a inpatient pulmonary rehabilitation program
  measured via Borg-scale at rest, during 6-minute walking distance, during constant work rate test at iso-time, during inspiratory muscle endurance capacity test

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Bavaria, Germany